CLINICAL TRIAL: NCT03842774
Title: Double Blind, Randomized Controlled Study to Evaluate the Efficacy and Safety of Extract of Gelidium Elegans
Brief Title: Efficacy and Safety of Extract of Gelidium Elegans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2017-0860
Record Dates: First submitted 2019-02-06; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): taken 3 tablets of Gelidium elegans extract (1000 mg/day) once a day for 12 weeks
  Interventions: Dietary Supplement: Exract of Gelidium elegans
- Control group (Placebo Comparator): taken 3 tablets of placebo once a day for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Exract of Gelidium elegans — Exract of Gelidium elegans will be given to the test group.
  Arms: Test group
Dietary Supplement: Placebo — Placebo supplement will be given to the test group.
  Arms: Control group

SUMMARY:
Extract of Gelidium elegans inhibits lipid differentiation, accumulation, and synthesis in vitro and in vivo. It has also anti-obesity effect by inhibiting weight gain and decreasing body fat. In a preliminary study of obese adults aged 20 years or older, the extracts of Gelidium elegans showed a tendency to decrease in body fat and visceral fat, and to increase lean body mass. Based on these results, we tried to confirm the effect of body weight and body fat reduction of Gelidium elegans extract in overweight and obese people.

ELIGIBILITY:
Inclusion Criteria:

* 1. Between the ages of 19 and 50
* 2. BMI is at or greater than 23 and less than 30 kg/m^2

Exclusion Criteria:

* 1. uncontrolled hypertension
* 2. uncontrolled diabetes
* 3. current serious cerebrovascular and cardiovascular disease

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-11-23 (Actual)

PRIMARY OUTCOMES:
change in body fat mass by DEXA after 12-week treatment | 12 week
change in visceral, subcutaneous, total fat area and ratio of visceral and subcutaneous fat area will be combined to report by Fat CT after 12-week treatment | 12 week

SECONDARY OUTCOMES:
change in body weight and body fat mass will be combined to report by Bio-impedance | 6 week
change in body weight and body fat mass will be combined to report by Bio-impedance | 12 week
change in waist circumference | 6 week
change in waist circumference | 12 week
change in hip circumference | 6 week
change in hip circumference | 12 week
change in ratio of waist and hip circumference | 6 week
change in ratio of waist and hip circumference | 12 week
body mass index | 6 week
body mass index | 12 week
change in lean body mass by DEXA | 6 week
change in lean body mass by DEXA | 12 week
change in laboratory test result of total cholesterol, HDL, LDL and triglyceride will be combined to report as lipid profile | 6 week
change in laboratory test result of total cholesterol, HDL, LDL and triglyceride will be combined to report as lipid profile | 12 week
change in laboratory test result of CRP | 6 week
change in laboratory test result of CRP | 12 week
change in laboratory test result of fasting insulin | 6 week
change in laboratory test result of fasting insulin | 12 week
change in HOMA-IR | 6 week
change in HOMA-IR | 12 week
change in HOMA-beta | 6 week
change in HOMA-beta | 12 week

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Family Medicine, Severance Hospital, College of Medicine, Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No